CLINICAL TRIAL: NCT01616251
Title: Acute Effect of Animal and Vegetable Protein Rich Meals With Comparable Dietary Fibers Content on Appetite Sensation and Energy Intake
Acronym: PAVA-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, Dr Med, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: B294
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Obesity
Keywords: Protein sources; Appetite; Dietary fibers; Meat; Egg; Legumes
MeSH Terms: conditions — Obesity | interventions — Energy Intake

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vegetable protein meal (Experimental): Vegetable protein meal based on legumes (3.6 MJ, 19E% protein, 28 g dietary fibers)
  Interventions: Other: Acute effect of animal and vegetable protein rich meals with comparable dietary fibers content on appetite sensation and energy intake
- Egg protein meal + fibers (Experimental): Protein meal based on eggs and added pea dietary fibers (3.6 MJ, 19E% protein, 28 g dietary fibers)
  Interventions: Other: Acute effect of animal and vegetable protein rich meals with comparable dietary fibers content on appetite sensation and energy intake
- Egg protein meal (Experimental): Protein meal based on egg without added dietary fibers (3.6 MJ, 19E% protein, 6 g dietary fibers)
  Interventions: Other: Acute effect of animal and vegetable protein rich meals with comparable dietary fibers content on appetite sensation and energy intake
- Meat protein meal + fibers (Experimental): Protein meal based on meat and added pea dietary fibers (3.6 MJ, 19E% protein, 29 g dietary fibers)
  Interventions: Other: Acute effect of animal and vegetable protein rich meals with comparable dietary fibers content on appetite sensation and energy intake

INTERVENTIONS:
Other: Acute effect of animal and vegetable protein rich meals with comparable dietary fibers content on appetite sensation and energy intake — 4-arm crossover study with the objective to examine if vegetable protein (beans and peas) can suppress subjective appetite (VAS and ad libitum EI) compared to isocaloric meals enriched with either red meat or egg with similar distribution of macronutrients and content of dietary fibers.

SUMMARY:
Background:

* New Nordic diet guidelines advocate a reduction in consumption of protein from animal sources such as beef and pork, due to environmental concerns.
* Instead, intake of protein from vegetable sources such as legumes and pulses should be increased.
* A previous study showed that a meal enriched with vegetable protein increased the subjective sensation of satiety and decreased hunger and ad libitum energy intake (EI) compared to animal protein.
* This study did, however, not document that vegetable protein per se is more satiating than animal protein as the vegetable meal had higher fiber content. Fiber is a likely confounder.
* The protein from egg is sparingly investigated in relation to appetite. Few studies have found that eggs have a high satiety index but further investigation is needed.

Objective:

- To examine if vegetable protein (beans and peas) can suppress subjective appetite (VAS and ad libitum energy intake) compared to isocaloric meals enriched with either red meat or egg with similar distribution of macronutrients and content of dietary fibers.

Design:

Single-blind randomized 4-way crossover meal study

Subjects:

33 young healthy men (Age: 18-50 years; BMI: 19-30 kg/m2). Expected completers: n=30.

End points:

1. Subjective appetite (VAS) (every 30 min for 3 hours)
2. Ad libitum EI (3 hours after lunch test meal)

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI: 18.5-30.0 kg/m2
* Weight stable (within +/- 3 kg) two months prior to study inclusion,
* Non-smoking
* Nonathletic (< 10 h hard physical activity)

Exclusion Criteria:

* BMI > 30 kg/m2
* Change in smoking status
* Daily or frequent use of medication that can affect appetite
* Suffering from metabolic diseases
* Suffering from psychiatric diseases
* Suffering from any other clinical condition, which would make the subject unfit to participate in the study
* alcohol and drug abuse
* food allergies or relevance for the test meals

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Ad libitum energy intake | Measured on 4 separate test days in a crossover design. Each test day is separated by >1 week. Assessed 180 min after each of the 4 test meals.
  180 min after each test meal an ad libitum meal of spaghetti bolognese is served, and the total energy intake is recorded.

SECONDARY OUTCOMES:
Acute 3-h changes from baseline in subjective appetite sensations using visual analogue scales | Measured on 4 separate test days in a crossover design. Each test day is separated by >1 week. On each test day appetite sensations are measured prior to the test meal (time 0) and 15, 30, 60, 90, 120, 150, 180 minutes post intake
  Assessment of subjective appetite sensations (visual analogue scales (VAS)) at time 0 (baseline - prior to the test meal) and at time 15, 30, 60, 90, 120, 150, 180 minutes post intake. Measured subjective appetite sensations of hunger, satiety, prospective consumption, fullness, composite appetite score and sensory desires to something sweet, salty, rich in fat, or meat/fish.
Rating of the organoleptic quality of the test meals | Measured on 4 separate test days in a crossover design. Each test separated by >1 week. On each test day after completion of the test meal subjects will rate the test meal
  After completion of the test meal the subjects will rate the organoleptic quality of the drink by visual analogue scales (VAS) in regard to appearance, smell, taste, after-taste, and general palatability.
Rating of the organoleptic quality of the ad libitum meal | Measured on 4 separate test days in a crossover design. Each test separated by >1 week. On each test day after completion of the ad libitum meal (approximately) time 15-20 minutes post intake) subjects will rate the ad libitum meal
  After completion of the adlibitum meal the subjects will rate the organoleptic quality of the meal by visual analogue scales (VAS) in regard to appearance, smell, taste, after-taste, and general palatability.
Subjective appetite sensations (visual analogue scales) after ad libitum meal | Measured on 4 separate test days in a crossover design. Each test separated by >1 week. After completion of the ad libitum meal subjects will rate their subjective sensation of appetite (approx 3.5-h post intake of test meal)
  After completion of the ad libitum meal the subjects will rate the subjective appetite sensations by visual analogue scales (VAS) in regard to sensation of hunger, satiety, prospective consumption, fullness, composite appetite score and sensory desires to eat something sweet, salty, rich in fat, or meat/fish.
Compensatory food intake (weighed dietary food record) | Measured on 4 separate test days in a crossover design. Each test separated by >1 week. Participants fill in a weighed food record from the time they complete the lunch until midnight.

CONTACTS AND LOCATIONS:
Overall Officials: Anne B Raben, PhD, Principal Investigator — Department of Human Nutrition, Faculty of Science, University of Copenhagen, Denmark
Locations (1):
- Department of Human Nutrition, Faculty of Science, University of Copenhagen, Frederiksberg, Denmark